CLINICAL TRIAL: NCT00152217
Title: Adjuvant Chemotherapy Trial of TS-1 for Gastric Cancer (ACTS-GC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91023038
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Cancer
Keywords: Stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; S 1 (combination); Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): TS-1 (S-1)
  Interventions: Drug: TS-1 (S-1)
- 2 (Other): Surgery alone
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: TS-1 (S-1) — 80 mg of oral S-1 per square meter of body-surface area per day was given for 4 weeks and no chemotherapy was given for the following 2 weeks
  Arms: 1
Procedure: Surgery — Stage II or III gastric cancer who underwent gastrectomy were assigned to surgery only
  Arms: 2

SUMMARY:
This controlled study is designed to evaluate the efficacy of TS-1 on survival compared with surgery alone. Patients will be randomly assigned to receive either surgery alone or surgery followed by treatment with TS-1 within 45 days after curative resection (curability A or B). To assess the efficacy, data on recurrence and survival will be collected from the time of enrollment until 5 years after surgery. To evaluate safety, data on adverse events will be collected from the time of enrollment until 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80
* Hematopoietic WBC ≥ 4,000/mm^3 Platelet ≥ 100,000/mm^3
* Hepatic AST and ALT ≤ 2.5 times upper limit of normal(ULN) Total bilirubin ≤ 1.5 mg/dL
* Renal Creatinine ≤ULN

Exclusion Criteria:

* Prior anticancer treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2001-09; Primary Completion 2007-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Relapse-free survival, adverse events | any time

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Sasako, MD, Principal Investigator — Department of Upper Gastrointestinal Surgery, Hyogo College of Medicine
Locations (1):
- National Cancer Center Hospital, 5-1-1, Tsukiji, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Result] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Derived] Ito S, Ohashi Y, Sasako M. Survival after recurrence in patients with gastric cancer who receive S-1 adjuvant chemotherapy: exploratory analysis of the ACTS-GC trial. BMC Cancer. 2018 Apr 20;18(1):449. doi: 10.1186/s12885-018-4341-6. PMID 29678146